CLINICAL TRIAL: NCT02115594
Title: A Phase 2, Randomized, Double-Blind, Multicenter Study of Fulvestrant With and Without Entinostat in Postmenopausal Women With Hormone Receptor-Positive Advanced Breast Cancer
Brief Title: Phase 2 Study of Fulvestrant With and Without Entinostat in Postmenopausal Women With ER+ Advanced Breast Cancer
Acronym: ENCORE305
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Internal decision
Sponsor: Syndax Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SNDX-275-0305
Record Dates: First submitted 2014-04-04; First posted 2014-04-16 (Estimated); Last update posted 2014-10-08 (Estimated); Status verified 2014-04

CONDITIONS: Breast Cancer
Keywords: metastatic breast cancer; estrogen receptor; Histone Deacetylase Inhibitors; Histone Deacetylases; HDAC inhibitors; selective estrogen receptor modulator; estrogen receptor modulator, selective; Estrogen receptor modulators, selective
MeSH Terms: conditions — Breast Neoplasms | interventions — Fulvestrant; entinostat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fulvestrant + Entinostat (Experimental): Arm A: Fulvestrant (500 mg on C1D1, C1D15, C2D1, and on Day 1 of each subsequent cycle) plus entinostat (5 mg PO once weekly)
  Interventions: Drug: Fulvestrant; Drug: Entinostat
- Fulvestrant + Placebo (Active Comparator): Arm B: Fulvestrant (500 mg on C1D1, C1D15, C2D1, and on Day 1 of each subsequent cycle) plus placebo (5 mg PO once weekly)
  Interventions: Drug: Fulvestrant; Drug: Placebo

INTERVENTIONS:
Drug: Fulvestrant
  Other Names: faslodex
Drug: Entinostat
  Arms: Fulvestrant + Entinostat
Drug: Placebo
  Arms: Fulvestrant + Placebo

SUMMARY:
Preclinical data has demonstrated that entinostat (SNDX-275) can enhance fulvestrant sensitivity in hormone receptor-positive breast cancer in animal models. The addition of entinostat to fulvestrant will provide clinical benefit to patients with locally advanced or metastatic breast when compared to fulvestrant plus placebo. Also, based on previous data, patients exposed to entinostat who demonstrate an elevated level of protein lysine acetylation will have an improved efficacy outcome.

DETAILED DESCRIPTION:
Entinostat (SNDX-275) inhibits mechanisms of resistance to hormone therapy in breast cancer (BC) cells, thereby prolonging sensitivity of the cells to fulvestrant. Preclinical data has demonstrated that entinostat can enhance fulvestrant sensitivity in hormone receptor-positive BC in animal models. Thus, it is hypothesized that the addition of entinostat to fulvestrant will provide clinical benefit to patients with locally advanced or metastatic BC when compared to fulvestrant plus placebo.

Preliminary data from Phase 2 Study SNDX-275-0301 suggest patients with higher levels of protein lysine acetylation who receive entinostat with exemestane potentially have improved clinical outcomes (e.g., PFS, OS) when compared to patients with lower levels of protein lysine acetylation. Thus, it is hypothesized that patients exposed to entinostat and who demonstrate an elevated level of protein lysine acetylation will have an improved efficacy outcome.

ELIGIBILITY:
Inclusion Criteria:

* Patient is a female who is: Postmenopausal OR Pre/perimenopausal and: Received at least one prior hormone therapy in combination with a luteinizing hormone-releasing hormone (LHRH) agonist prior to study entry. Initiated on an LHRH agonist at least 28 days prior to study entry. Demonstrated ovarian estradiol suppression, defined as an estradiol level within postmenopausal ranges per institutional guidelines, within 28 days immediately prior to study entry
* Patient has histologically or cytologically confirmed ER+ and/or progesterone receptor-positive (PR+) BC at initial diagnosis or on subsequent biopsy. With regard to hormone receptor status, staining of ≥1% cells is considered positive. Receptor status may have been determined at any time prior to randomization and from any site (i.e., primary, recurrent, or metastatic)
* Patient experienced PD within 28 days before initiating study treatment and has been deemed eligible for treatment with fulvestrant
* Patient has evidence of locally advanced or metastatic disease, based on imaging studies (bone scan, CT, MRI) within 28 days before initiating study treatment
* Patient completed any prior radiotherapy ≥2 weeks prior to receiving the first dose of study treatment and has recovered from any radiation-related toxicity
* Patient may have received 1 prior chemotherapy regimen for metastatic disease provided treatment was completed ≥3 weeks prior to randomization. Prior chemotherapy in the adjuvant or neoadjuvant setting is also allowed
* Patient is willing and able to provide or assist study personnel in accessing slides from prior biopsies
* Patient has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Patient has the following laboratory parameters: a. Hemoglobin (Hgb) ≥9.0 g/dL; unsupported platelet count ≥100×10P9P/L; and absolute neutrophil count (ANC) ≥1.5×10P9P/L without the use of hematopoietic growth factors; b. Creatinine ≤2.0 mg/dL; c. Total bilirubin <1.5 x institutional upper limit normal (≤3 mg/dL in case of Gilbert's syndrome); d. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2 x institutional upper limit of normal; unless elevation is due to metastatic disease to the liver, in which case ALT and AST must be within 5.0 x institutional upper limit of normal
* Patient is able to swallow tablets
* Patient is able to understand and give written informed consent and comply with study procedures

Exclusion Criteria:

* Patient has rapidly progressive or life-threatening metastases (visceral crisis)
* Patient has HER2-positive (HER2+) disease, as defined by the 2013 American Society of Clinical Oncology (ASCO)/College of American Pathologists (CAP) recommendations for HER2 testing in BC (see http://www.asco.org/quality-guidelines/recommendations-human-epidermal-growth-factor-receptor-2-testing-breast-cancer), or has unknown HER2 status
* Patient previously received treatment with entinostat or any other HDAC inhibitor, including valproic acid
* Patient has had previous treatment with fulvestrant or other selective estrogen receptor down-regulator (SERD) in the metastatic setting; such treatment may have been given in the adjuvant setting
* Patient has an allergy to benzamide or inactive components of the study drug
* Patient has a history of allergies to any active or inactive ingredients of fulvestrant
* Patient has a concomitant medical condition that precludes adequate study treatment compliance or assessment, or increases patient risk, in the opinion of the Investigator, such as but not limited to:

  1. Myocardial infarction or arterial thromboembolic event within 6 months prior to Baseline or severe or unstable angina, New York Heart Association (NYHA) Class III or IV disease (see Appendix 2), or a QTc interval >470 msec.
  2. Uncontrolled heart failure or hypertension, uncontrolled diabetes mellitus, or uncontrolled systemic infection
  3. Another active cancer (excluding adequately treated basal cell carcinoma or cervical intraepithelial neoplasia [CIN] / cervical carcinoma in situ or melanoma in situ). Prior history of other cancer is allowed, as long as there is no active disease within the prior 5 years
* Patient is currently receiving treatment with any agent listed on the prohibited medication list such as valproic acid or other systemic cancer agents
* Patient initiated oral bisphosphonates within 7 days prior to study drug
* Patient has moderate or severe hepatic impairment (i.e., Child-Pugh score B or C)
* Patient has brain or leptomeningeal metastases

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-04; Primary Completion 2015-12 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | From date of randomization until the date of 1st documented progression or date of death from any cause, whichever occurs first, assessed for up to 48 months
  Radiological disease assessments

SECONDARY OUTCOMES:
Objective Response Rate (CR or PR) | From date of randomization until the date of 1st documented progression or date of death from any cause, whichever occurs first, for up to 48 months
  Radiological disease assessments
Clinical Benefit Rate (CR, PR, or SD for greater than or equal to 6 months from randomization) | From the date of randomization until the date of 1st documented progression or date of death, from any cause, whichever occurs first, assessed for up to 48 months
  Radiological disease assessments
Overall Survival | From the date of randomization until date of death, assessed for up to 48 months
Clinical review of safety parameters (AEs, lab values) | From date of randomization until 30 days post the date of study treatment discontinuation
Percent change from baseline in blood protein lysine acetylation measures | From the baseline visit through the 1st 15 days of study treatment
Concentrations of entinostat measured in plasma (PK) | From the baseline visit through the 1st 15 days of study treatment

OTHER OUTCOMES:
Analysis of biopsy tumor tissue (fresh optional, archival required) | Screening (fresh tissue) and post 1st dose, between Days 15-18 of study treatment
  molecular classification of breast cancer (BC) subtypes, DNA methylation, e-cadherin levels, protein lysine acetylation levels, and changes in proteins associated with estrogen signaling and fulvestrant resistance

CONTACTS AND LOCATIONS:
Overall Officials: Denise Yardley, MD, Principal Investigator — Tennessee Oncology / Sarah Cannon
Locations (1):
- Tennessee Oncololgy, Nashville, Tennessee, United States